CLINICAL TRIAL: NCT06209099
Title: Organ Preservation First Strategy and Intentional Watch and Wait for MRI Defined Low-risk Rectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Lin Wang, Unit III & Ostomy Service, Gastrointestinal Cancer Center, Peking University Cancer Hospital & Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKUCH-R08
Record Dates: First submitted 2024-01-06; First posted 2024-01-17 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Rectal Cancer
Keywords: organ preservation, chemoradiotherapy, neoadjuvant, rectal cancer, watch and wait
MeSH Terms: conditions — Rectal Neoplasms | interventions — Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A: Nonoperative Management (Experimental): Patients who achieve Clinical complete response (cCR) or near-cCR when restaged at 16 weeks following IMRT plus consolidation CapeOX.
  Interventions: Procedure: Nonoperative Management (NOM)
- Group B: Local Excision (Experimental): Patients with near-cCR or residual tumor ≤ycT2N0 when reassessed at 16 weeks following IMRT plus consolidation CapeOX; or Patients with regrowth ≤ycT2N0 when reassessed during surveillance in NOM;
  Interventions: Procedure: Local Excision (LE)
- Group C: Total Mesorectal Excision (Experimental): Patients with residual tumor >ycT2N0 when restaged at 16 weeks following IMRT plus consolidation CapeOX.
  or Patients with regrowth >ycT2N0 when reassessed during surveillance in NOM; or Patients with any high-risk pathological factors following local excision (LE)
  Interventions: Procedure: Total Mesorectal Excision (TME)

INTERVENTIONS:
Procedure: Nonoperative Management (NOM) — Drug: Oxaliplatin (OXA) Drug: Capecitabine (CAPE) Radiation: intensity modulated radiotherapy (IMRT) Behavioral: DRE-Endoscopy-MRI-CEA Procedure: Nonoperative Management (NOM)
  Arms: Group A: Nonoperative Management
Procedure: Local Excision (LE) — Drug: Oxaliplatin (OXA) Drug: Capecitabine (CAPE) Radiation: intensity modulated radiotherapy (IMRT) Behavioral: DRE-Endoscopy-MRI-CEA Procedure: Local Excision (LE)
  Arms: Group B: Local Excision
Procedure: Total Mesorectal Excision (TME) — Drug: Oxaliplatin (OXA) Drug: Capecitabine (CAPE) Radiation: intensity modulated radiotherapy (IMRT) Behavioral: DRE-Endoscopy-MRI-CEA Procedure: Total Mesorectal Excision (TME)
  Arms: Group C: Total Mesorectal Excision

SUMMARY:
The goal of this clinical trial is to test the safety and efficacy of local excision (LE) or non-operative management (NOM) in patients with MRI defined low-risk rectal cancer following neoadjuvant intensity modulated radiotherapy with concurrent capecitabine plus consolidation CapeOX. The main questions it aims to answer are:

1. What is the organ-preservation rate (OPR) after in patients with MRI defined low-risk rectal cancer following neoadjuvant intensity modulated radiotherapy with concurrent capecitabine plus consolidation CapeOX?
2. Is LE or NOM safe and effective in patients with MRI defined low-risk rectal cancer following neoadjuvant intensity modulated radiotherapy with concurrent capecitabine plus consolidation CapeOX? Participants will receive radical surgery, LE, or NOM based on the response of neoadjuvant intensity modulated radiotherapy with concurrent capecitabine plus consolidation CapeOX in patients with MRI defined low-risk rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤85 years
* ECOG Performance status 0-1
* Histologically confirmed diagnosis of adenocarcinoma of the rectum, with tumor differentiation Grade 1-3
* The distance from down verge of tumor to anal-rectal junction (ARJ) ≤4cm based on MRI, or ≤8 cm based on sigmoidoscopy
* Clinical Stage T2 or T3a or T3b and EMVI (-) and MRF (-) and extra-mesorectal metastatic lymph node (-) based on MRI
* The maximum diameter of the tumor is ≤4cm or the circumferential invasion range is less than 1/3 of the intestinal circumference
* No evidence of distant metastases
* No prior pelvic radiation therapy
* No prior chemotherapy or surgery for rectal cancer
* No active infections requiring systemic antibiotic treatment
* ANC > 1.5 cells/mm3, HGB > 10.0 g/dL, PLT > 100,000/mm3, total bilirubin ≤ 1.5 x ULN, AST≤ 3 x ULN, ALT ≤ 4 x ULN
* Patients must read, agree to, and sign a statement of Informed Consent prior to participation in this study.

Exclusion Criteria:

* Recurrent rectal cancer
* Primary unresectable rectal cancer. A tumor is considered unresectable when invading adjacent organs and an en-bloc resection will not achieve negative margins
* Creatinine level greater than 1.5 times the upper limit of normal
* Patients who have received prior pelvic radiotherapy
* Patients who are unable to undergo an MRI
* Patients with a history of a prior malignancy within the past 5 years, except for well treated basal cell cancer, squamous cell skin cancer, breast cancer, thyroid cancer or small renal cancer, and with DFS >5 years
* Patients with a history of any arterial thrombotic event within the past 6 months. This includes angina (stable or unstable), MI, TIA, or CVA
* Other anticancer or experimental therapy
* Women who are pregnant or breast-feeding
* Patients with any other concurrent medical or psychiatric condition or disease which would make them inappropriate candidates for entry into this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Organ-preservation rate | Three years
  The rate of organ preservation will be defined as the percentage of patients who achieve cCR or near-cCR after neoadjuvant treatment followed by local excision or non-operative management (NOM). The time of organ preservation will be measured from the initiation of treatment.

SECONDARY OUTCOMES:
Rate of non-regrowth disease-free survival (NR-DFS) | Three years
  NR-DFS will be defined as the length of time after treatment until death (any cause), tumor relapse including local pelvic recurrence following TME or local resection and any distant metastasis during or after treatment. Surgical salvageable local regrowth occurs in non-operative management will not be defined as tumor relapse.
Stoma-free survival | Three years
  Stoma-free survival will be defined as the length of time in which patients live with a temporary or permanent stoma and be measured from the initiation of treatment. Events for stoma-free survival are temporary or permanent stoma or death (any cause). Temporary ileostomy-free survival or colostomy-free survival will also be calculated.
Major adverse events | Three years
  Adverse events will be graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Haidian District, China

IPD SHARING:
Plan to Share IPD: No